CLINICAL TRIAL: NCT03950297
Title: A First-in-Human, Open-label, Phase 1 Dose-Escalation Study of 609A in Subjects With Locally Advanced / Metastatic Solid Tumors
Brief Title: Phase 1, First in Human, Open-Label, Dose-Escalation Study of 609A
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunshine Guojian Pharmaceutical (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SSGJ-609-UND-US-I-01
Record Dates: First submitted 2019-05-13; First posted 2019-05-15 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2019-05

CONDITIONS: Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 609A group (Experimental): Dose escalation will be conducted using a traditional 3+3 design. Dose Escalation Level cohort 1. Dose 1 mg/kg, Q3W, IV. Subjects 3-6; Dose Escalation Level cohort 2. Dose 3 mg/kg, Q3W, IV. Subjects 3-6; Dose Escalation Level cohort 3. Dose 200mg, Q3W, IV. Subjects 3-6; Dose Escalation Level cohort 4. Dose 10 mg/kg, Q3W, IV. Subjects 3-6;
  Interventions: Drug: 609A

INTERVENTIONS:
Drug: 609A — 609A is a recombinant anti-PD-1 humanized IgG4 kappa antibody that targets the human PD-1

SUMMARY:
Phase 1, First in Human, Open-Label, Dose-Escalation Study of 609A in the Patients with Locally advanced/Metastatic Solid Tumors

DETAILED DESCRIPTION:
This is a first-in-human (FIH), open-label, phase 1 dose-escalation study of 609A, a recombinant monoclonal anti-PD-1 antibody product, in subjects with Locally advanced/Metastatic Solid Tumors, who must have received, or be intolerant to all available approved or standard therapies known to confirm clinical benefit, or for whom no standard therapy exits.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all the following inclusion criteria to be eligible for participation in this study:

* Able to understand and willing to sign the Informed Consent Form(ICF).
* Male or female ≥ 18years.
* Subjects with histologically or cytologically confirmed advanced-stage or metastatic tumor must have received, or be intolerant to all available approved or standard therapies known to confirmed clinical benefit, or for whom standard therapy does not exist.
* Must have adequate organ function, prior to start of 609A, including the following:

  1. Bone marrow reserve: absolute neutrophil count (ANC) ≥ 1.0 ×109/L; platelet count≥ 100 × 109/L; hemoglobin ≥ 9 g/dL or ≥ 5.6 mmol/L;
  2. Hepatic: total bilirubin ≤ 1.5 times the upper limit of normal (ULN), aspartate transaminase (AST) and/or alanine aminotransferase (ALT) ≤ 3 × ULN (≤5 × ULN if with liverinvolvement)
  3. Renal: serum creatinine ≤1.5 times the ULN or estimated creatinineclearance

     ≥50mL/min (Cockroft and Gault formula [http://www.mdcalc.com/creatinine-clearance-cockcroft-gault-equation/]).
  4. Coagulation tests INR≤ 2 (Exception: INR 2 to ≤ 3 is acceptable for subjects onWarfarin anticoagulation), activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN
* Regarding prior anti-tumortherapy:

  1. Subjects who have received any anticancer drugs approved or investigational, including chemotherapy, immune therapy, hormonal therapy (Exceptions: hormone-replacement therapy, testosterone or oral contraceptives), biologic therapy, must have stopped treatment at least 3 weeks, or five half-lives, whichever is shorter, before first dose of 609A.
  2. Generalized radiation therapy must have stopped 3 weeks before first dose of 609A, or local radiotherapy or radiation therapy for bone metastases must have stopped 2 weeks before first dose of 609A. No therapeutic radiopharmaceuticals are taken within 8 weeks before first dose of 609A.
  3. Subjects who have received prior immunotherapies targeting T cell stimulation such as (e.g. anti-PD-1, anti- PD-L1 or anti-CTLA-4) must have stopped treatment for at least 4 weeks before first dose of 609A.
* Female patient with fertility or male patient whose partner has fertility should use one or more contraceptive methods for contraception from the screening period to five half-lives after the last treatment. These measures include, but are not limited to, oral or implantable injections of hormonal contraceptives; intrauterine birth control ring or placement of intrauterine system (IUS) hormone-releasing intrauterine device; or use of barrier methods such as condoms or septum and spermicide products. Women of childbearing potential must have a negative pregnancy test ≤ 72 hours prior to the first dose of study drug.

Postmenopausal women must have been amenorrhoeic for at least 12 months to be considered of non-childbearing potential.

* According to RECIST1.1, the subject should have an assessable lesion (target lesion or non- target lesion)
* According to RECIST1.1, the subject should have an assessable lesion (target lesion or non- target lesion) ECOG score 0, 1 or 2 point.

Exclusion Criteria:

* Subjects who meet any of the following criteria cannot be enrolled: Life expectancy < 3 months.
* Any remaining AEs > grade 1 from prior anti-tumor treatment as per CTCAE v5. 0, with exception of the residual hair loss;
* Any remaining AEs > grade 1 from prior anti-tumor treatment as per CTCAE v5. 0, with exception of the residual hair loss; Any involvement of CNS excluded except: Based on screening brain magnetic resonance imaging (MRI), patients must have one of the following:

  1. No evidence of brain metastases or has to be clinically stable for at least 4 weeks
  2. Untreated brain metastases not needing immediate localtherapy
* Pregnant or nursing females
* Subjects who have had major surgery within the 21-days from the screening;
* Subjects with history of interstitial lung disease or idiopathic pulmonary fibrosis or unresolved active or chronic inflammatory pulmonary disease are excluded. Subjects with a history of radiation pneumonitis which has resolved areeligible.
* HIV infection.
* Active hepatitis B or C. HBV carriers without active disease (HBV DNA titer< 1000 cps/mL or 200 IU/mL) or cured Hepatitis C (negative HCV RNA test) may been rolled.
* History of primary immunodeficiency, stem cell or organ transplant, or previous clinical diagnosis of tuberculosisdisease.
* History of life-threatening hypersensitivity or known to be allergic to protein drugs or recombinant proteins or excipients in 609A drug formulation.
* Acute or chronic uncontrolled renal disease, pancreatitis or liver disease (per investigator assessment).
* Subjects with any type of primary immunodeficiencies will be excluded from thestudy.
* Subjects with condition requiring systemic treatment with either corticosteroids (>15 mg/day prednisone or equivalent) or other immunosuppressive medications within 14 days before the planned first dose of study drug. Inhaled or topical steroids, and adrenal replacement steroid doses ≤ 10 mg daily prednisone equivalent are permitted in the absence of activeautoimmune disease. Ophthalmologic, nasal and intra-articular injections of steroids areacceptable.
* Subjects who experienced immunotherapy-related adverse events (irAE) grade ≥ 3, or who had to discontinue prior anti-PD-1, anti-PD-L1, or CTL4 treatment due to irAEs of any grade.
* Severe or uncontrolled cardiac disease requiring treatment, congestive heart failure NYHA III or IV, unstable angina pectoris even if medically controlled, history of myocardial infarction during the last 6 months, ECG QTcF (Fridericia)≥450 msec for male or QTcF (Fridericia)≥470 msec for female, serious arrhythmias requiring medication (with exception of atrial fibrillation or paroxysmal supraventricular tachycardia).
* Hypertension (defined as sustained systolic blood pressure> 160 mm Hg and / or post- diastolic blood pressure with antihypertensive drugs> 100 mmHg;
* Any other serious underlying medical (e.g. uncontrolled diabetes mellitus, active uncontrolled infection, active gastric ulcer, uncontrolled seizures, cerebrovascular incidents, gastrointestinal bleeding, severe signs and symptoms of clotting disorders), psychiatric, psychological, familial or geographical condition that, in the judgment of the investigator, may interfere with the planned staging, treatment and follow-up, affect subject compliance or place the subject at high risk from treatment-related complications.
* Has received a live and attenuated vaccine within 28 days prior to the first dose of study drug.
* Patients who had received treatment with any herbal or alternative therapies or Chinese prepared medicine within 7 days prior to the first dose of the studydrug.
* Subjects with active autoimmune diseases or history of autoimmune diseases should be excluded; these include but are not limited to subjects with a history of immune related neurologic disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain- Barre syndrome, myasthenia gravis, systemic lupus erythematosus (SLE), connective tissue diseases, scleroderma, inflammatory bowel disease including Crohn's disease and ulcerative colitis, hepatitis, toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome, or antiphospholipidsyndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-10-24 (Estimated); Study Completion 2022-05-24 (Estimated)

PRIMARY OUTCOMES:
Treatment-Emergent Adverse Events | for 90 Days
  To monitor adverse events (AEs) per the NCI CTCAE 5.0.
The MTD | for 90 Days
  Maximum Tolerated Dose, if any, and RP2D (s) for 609A will be determined.

SECONDARY OUTCOMES:
AUC | for 90 Days
  Area Under the Curve of 609A
Cmax | for 90 Days
  Maximum Plasma Concentration of 609A
t½ | for 90 Days
  Half life of 609A in blood
CL | for 90 Days
  Plasma clearance of 609A
ORR | for 1 Year
  the rate of completely response [CR] and partial response [PR] patients
DCR | for 1 Year
  disease control rates of the patients with 609A
PFS | for 1 Year
  Progression-free survival of the patients with 609A
DOR | for 1 Year
  Duration of response of the patients with 609A
OS | for 1 Year
  overall survival of the patients with 609A
Immunogenicity | for 1 Year
  the presence of anti-609A antibody will be assessed

CONTACTS AND LOCATIONS:
Locations (1):
- NEXT Oncology Business Office, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No